CLINICAL TRIAL: NCT02655770
Title: Influence of Liraglutide on Diastolic Cardiac Function and Myocardial Perfusion as Determined by Magnetic Resonance Imaging in Patients With Type 2 Diabetes: a Double-blind Randomized Parallel-group Trial
Brief Title: Effect of Liraglutide on Diastolic Dysfunction on Cardiac MRI in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Slagelse Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Annemie Stege Bojer, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-000410-22; 2015-000410-22 (EudraCT Number)
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus Type 2; Diastolic Dysfunction; Cardiac MRI; Myocardial Perfusion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide arm (Active Comparator): Patients will be treated with liraglutide (up to 1.8 mg s.c. once daily). Total treatment period will be 18 weeks.
  Interventions: Drug: Liraglutide
- Placebo arm (Placebo Comparator): Patients will be treated with placebo (up to equal to 1.8 mg drug dose s.c. once daily). Total treatment period will be 18 weeks. The study will be placebo-controlled with placebo as an add-on to conventional diabetes treatment. Thus, no patient will receive a sub-standard treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Liraglutide arm
Drug: Placebo
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to determine whether liraglutide a GLP-1 analogue are effective in the treatment of diastolic dysfunction in type 2 diabetes patients analyzed by cardiac MRI. Secondary if the treatment has any effect on the perfusion of the heart on a cardiac-MRI.

DETAILED DESCRIPTION:
Aim: To test if treatment with liraglutide a GLP-1 analogue in 18 weeks improves diastolic performance in type 2 diabetes (DM2) patients with diastolic dysfunction, compared to placebo. Furthermore, analyzing cardiac MRI indices of fibrosis and the effect on myocardial perfusion.

The investigators find that especially diastolic dysfunction is of interest, because it is highly overrepresented in DM2 patients and no treatment exists. Glucagon-like peptide 1 analogue could be a possible treatment agent, by increasing the energy level in the myocardium. No previous study has tested the effect of treatment with a glucagon-like peptide 1 analogue on diastolic dysfunction.

Design: A randomised double-blinded placebo-controlled clinical trial. Sample size: 40 patients, 20 in each group. The superior inter-study reproducibility results in considerably lower calculated sample sizes (reductions of 55% to 93%) required by cardiac MR compared with echocardiography to show clinically relevant changes. Power calculations show that only 30 patients are needed form our primary outcome, to allow for dropouts the investigators have chosen to include 40 patients.

Intervention: After randomization, patients will be treated with placebo or liraglutide (up to 1.8 mg s.c. once daily). Total treatment period will be 18 weeks. A cardiac MRI scan and an echocardiography will be preformed at baseline and after 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient fully capable of informed consent
* Informed consent
* Age 18-80 years (both years inclusive)
* T2DM diagnosed at least 3 months prior to visit 0
* NYHA class I-III at visit 0
* E/e* ≥ 9 or e* (lateral) ≤10 cm/sec, or both
* LVEF > 50%
* LVEDV/BSA < 97 ml/m2
* Stable on heart medication for 6 weeks prior to randomisation
* Stable on antidiabetic treatment for 30 days prior to randomisation
* T2DM must be either treated with one or more oral anti-diabetic drugs or treated with human NPH-insulin or long-acting insulin analogue, alone or in combination with oral drugs

Exclusion Criteria:

* Lack of consent.
* NYHA class IV
* Type 1 diabetes mellitus
* Incretin-based therapy (GLP-1 receptor agonists; exenatide, liraglutide or other and DPP-IV inhibitors) within 30 days prior to randomisation (visit 1)
* Glitazon therapy within 30 days prior to randomisation (visit 1)
* Hypertension with inadequate blood pressure control: Systolic blood pressure > 140 mmHg and/or diastolic blood pressure >85 mmHg*
* Supine systolic blood pressure <85 mmHg measured at visit 0
* Significant valvular heart disease
* Hypertrophic cardiomyopathy, ARVC/D, non-compaction or amyloidosis
* Myocardial infarction, unstable angina, angina on exertion (≥CCS class 2) or coronary revascularization within 3 months prior to randomisation (visit 1)
* Hospitalisation due to incompensated heart disease within 30 days to randomisation (visit 1)
* HbA1c >10% at visit 0
* eGFR< 60 ml/min/1,73 m2 at visit 0
* Liver disease with aspartate aminotransferase/alanine aminotransferase >3 times upper limit of normal measured at visit 0**
* Hypokalaemia (P-potassium <3.5 mmol/L) or hyperkalaemia (P-potassium >5.5 mmol/L) measured at visit 0**
* Anaemia (haemoglobin <6.5 mmol/L) measured at visit 0**
* Conditions that may be associated with changes in markers of fibroses or collagen turnover (eg. on-going or active rheumatological disease requiring anti-inflammatory agents, immunosuppression, pulmonary fibrosis, active cancer)
* Prolonged use (> 2 weeks) of glucocorticoids or NSAIDs within 2 weeks prior to visit 0
* Women of childbearing potential who are not on acceptable contraception. See below.
* Pregnant or breastfeeding women
* Cancer (except basal cell skin cancer or squamous cell skin cancer) unless complete remission for ≥ 5 years
* Alcohol/drug abuse
* Chronic or previous acute pancreatitis
* History of thyroid adenoma or carcinoma
* Inflammatory bowel disease
* Clinical signs of diabetic gastroparesis
* ICD/pacemaker or other contraindications to MRI scan
* Severe claustrophobia
* Atrial fibrillation
* Contraindications to glycopyrrolate: closed-angle glaucoma, prostate hyperplasia, tachycardia, bladder atony, cardia insufficiency, non-congenital pylorus stenosis and gastroparesis
* Known or suspected hypersensitivity to trial product or related products
* Current participation in any other clinical intervention trial
* Receipt of an investigational drug with 30 days prior to visit 0
* Other concominant disease or treatment that according to investigator's assessment makes the patient unsuitable for participation in the study

  * Measured twice at visit 0. In case of elevation, an ambulatory (24-hour) blood pressure will be performed, and the result of this will be conclusive

    * Measured at visit 0 with the possibility of one repeat analysis within a week, and the last measured value will be conclusive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in diastolic properties as assessed by CMR. | Measured in week 18 and compared to baseline.
  LA passive emptying fraction (%) (before and after glycopyrolate)
Change in diastolic properties as assessed by CMR. | Measured in week 18 and compared to baseline.
  LV peak filling rate (ml/s) (before and after glycopyrolate)

SECONDARY OUTCOMES:
MRI indices of myocardial perfusion | Measured in week 18 and compared to baseline.
Echocardiographic indices of diastolic dysfunction | Measured in week 18 and compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vejlstrup, MD, Med.Sc.D, Study Director — Rigshospitalet, Denmark
Locations (1):
- The department of cardiology, Rigshospitalet Denmark, Copenhagen Ø, Denmark

REFERENCES:
- [Background] Kannel WB, Hjortland M, Castelli WP. Role of diabetes in congestive heart failure: the Framingham study. Am J Cardiol. 1974 Jul;34(1):29-34. doi: 10.1016/0002-9149(74)90089-7. No abstract available. PMID 4835750
- [Background] Factor SM, Okun EM, Minase T. Capillary microaneurysms in the human diabetic heart. N Engl J Med. 1980 Feb 14;302(7):384-8. doi: 10.1056/NEJM198002143020706. No abstract available. PMID 7351930
- [Background] Nitenberg A, Paycha F, Ledoux S, Sachs R, Attali JR, Valensi P. Coronary artery responses to physiological stimuli are improved by deferoxamine but not by L-arginine in non-insulin-dependent diabetic patients with angiographically normal coronary arteries and no other risk factors. Circulation. 1998 Mar 3;97(8):736-43. doi: 10.1161/01.cir.97.8.736. PMID 9498536
- [Background] Rodrigues B, McNeill JH. The diabetic heart: metabolic causes for the development of a cardiomyopathy. Cardiovasc Res. 1992 Oct;26(10):913-22. doi: 10.1093/cvr/26.10.913. No abstract available. PMID 1486584
- [Background] van Heerebeek L, Hamdani N, Handoko ML, Falcao-Pires I, Musters RJ, Kupreishvili K, Ijsselmuiden AJ, Schalkwijk CG, Bronzwaer JG, Diamant M, Borbely A, van der Velden J, Stienen GJ, Laarman GJ, Niessen HW, Paulus WJ. Diastolic stiffness of the failing diabetic heart: importance of fibrosis, advanced glycation end products, and myocyte resting tension. Circulation. 2008 Jan 1;117(1):43-51. doi: 10.1161/CIRCULATIONAHA.107.728550. Epub 2007 Dec 10. PMID 18071071
- [Background] From AM, Scott CG, Chen HH. The development of heart failure in patients with diabetes mellitus and pre-clinical diastolic dysfunction a population-based study. J Am Coll Cardiol. 2010 Jan 26;55(4):300-5. doi: 10.1016/j.jacc.2009.12.003. PMID 20117433
- [Background] Yancy CW, Lopatin M, Stevenson LW, De Marco T, Fonarow GC; ADHERE Scientific Advisory Committee and Investigators. Clinical presentation, management, and in-hospital outcomes of patients admitted with acute decompensated heart failure with preserved systolic function: a report from the Acute Decompensated Heart Failure National Registry (ADHERE) Database. J Am Coll Cardiol. 2006 Jan 3;47(1):76-84. doi: 10.1016/j.jacc.2005.09.022. Epub 2005 Dec 15. PMID 16386668
- [Background] Bhashyam S, Fields AV, Patterson B, Testani JM, Chen L, Shen YT, Shannon RP. Glucagon-like peptide-1 increases myocardial glucose uptake via p38alpha MAP kinase-mediated, nitric oxide-dependent mechanisms in conscious dogs with dilated cardiomyopathy. Circ Heart Fail. 2010 Jul;3(4):512-21. doi: 10.1161/CIRCHEARTFAILURE.109.900282. Epub 2010 May 13. PMID 20466848
- [Background] Thrainsdottir I, Malmberg K, Olsson A, Gutniak M, Ryden L. Initial experience with GLP-1 treatment on metabolic control and myocardial function in patients with type 2 diabetes mellitus and heart failure. Diab Vasc Dis Res. 2004 May;1(1):40-3. doi: 10.3132/dvdr.2004.005. PMID 16305055
- [Background] Nathanson D, Ullman B, Lofstrom U, Hedman A, Frick M, Sjoholm A, Nystrom T. Effects of intravenous exenatide in type 2 diabetic patients with congestive heart failure: a double-blind, randomised controlled clinical trial of efficacy and safety. Diabetologia. 2012 Apr;55(4):926-35. doi: 10.1007/s00125-011-2440-x. Epub 2012 Jan 13. PMID 22246377